CLINICAL TRIAL: NCT00053950
Title: A Phase I Study of High-dose Pyrazoloacridine (PZA) (NSC 366140) Supported With Autologous Hematopoietic Stem Cell Rescue in Children With Recurrent or Resistant Neuroblastoma (IND # 36325)
Brief Title: Pyrazoloacridine and Stem Cell or Bone Marrow Transplantation in Treating Young Patients With High-Risk Neuroblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03166; NANT N2002-01; P01CA081403 (NIH); CHLA-NANT-N2002-01; CDR0000269644
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Disseminated Neuroblastoma; Recurrent Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — NSC 366140; Filgrastim; Granulocyte Colony-Stimulating Factor; Bone Marrow Transplantation; Transplantation; Peripheral Blood Stem Cell Transplantation

ARMS (2):
- Cohort I (Experimental): Groups of 3-6 patients receive escalating doses of PZA at a fixed infusion time until the MTD is determined. In both cohorts the MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Patients receive G-CSF IV or subcutaneously beginning on day 4 and continuing until blood counts recover. Patients also undergo reinfusion of stem cells over 15-30 minutes on day 4 as needed per protocol.
  Interventions: Drug: pyrazoloacridine; Biological: filgrastim; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis; Other: pharmacological study
- Cohort II (Experimental): Groups of 3-6 patients receive PZA at the dose/hour established in cohort I at escalating infusion times until another MTD is determined. In both cohorts the MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Patients receive G-CSF IV or subcutaneously beginning on day 4 and continuing until blood counts recover. Patients also undergo reinfusion of stem cells over 15-30 minutes on day 4 as needed per protocol.
  Interventions: Drug: pyrazoloacridine; Biological: filgrastim; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: pyrazoloacridine — Given IV
  Other Names: PZA
Biological: filgrastim — Given IV or SC
  Other Names: G-CSF; Neupogen
Procedure: autologous bone marrow transplantation — Undergo autologous bone marrow transplantation
  Other Names: ABMT; bone marrow transplantation, autologous; transplantation, autologous bone marrow
Procedure: peripheral blood stem cell transplantation — Undergo peripheral blood stem cell transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of pyrazoloacridine given together with peripheral stem cell or bone marrow transplantation in treating young patients with high-risk neuroblastoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell or bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of PZA given as a single prolonged infusion (>= 6 hours) with autologous hematopoietic stem cell (aHSC) support to children with high risk neuroblastoma with recurrent or refractory disease.

II. To determine the dose limiting toxicity (DLT) of PZA given on this schedule.

III. To characterize the pharmacokinetics of PZA given on this schedule.

SECONDARY OBJECTIVES:

I. To obtain preliminary data on the antitumor activity of PZA within the confines of a Phase I study.

II. To determine the TP53 mutation status of tumor cells in bone marrow if > 10% are present; to evaluate expression of p53 and MDM2 proteins by flow cytometry if >= 0.1% to < 10% are present at study entry.

OUTLINE: This is a two-stage, dose-escalation study.

Patients without adequate cryopreserved hematopoietic stem cells undergo peripheral blood stem cell harvest or bone marrow harvest for autologous stem cells at least 2 weeks before study therapy.

Patients receive high-dose pyrazoloacridine (PZA) IV on day 0.

Cohort 1: Groups of 3-6 patients receive escalating doses of PZA at a fixed infusion time until the maximum tolerated dose (MTD) is determined.

Cohort 2: Groups of 3-6 patients receive PZA at the dose/hour established in cohort I at escalating infusion times until another MTD is determined.

In both cohorts the MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients receive filgrastim (G-CSF) IV or subcutaneously beginning on day 4 and continuing until blood counts recover. Patients also undergo reinfusion of stem cells over 15-30 minutes on day 4 as needed per protocol.

Patients are followed at days 28-35, every 3 months for 3 years, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of neuroblastoma (ICD-O morphology 9500/3) verified by histology and/or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites
* Patients must meet one of the two following disease status criteria to enter on study;

  * Current or prior progressive disease (PD) by INRC criteria
  * Either mixed response (MR) or no response (NR) by INRC criteria following completion of minimum of 4 courses of induction therapy
* Patients meeting disease status criteria in either category A or B must also have at least one of the following sites of disease present to enter on study:

  * At least one tumor lesion on CT or MRI scan that is >= 20mm in at least one dimension (spiral CT lesion must be >= 10mm in at least one dimension)
  * MIBG scan with positive uptake at a minimum of one site
  * Bone marrow disease documented by standard histology of bilateral bone marrow aspirate and biopsy specimens
* Patients > 16 years of age: Karnofsky >= 50%; Patients =< 16 years of age: Lansky >= 50%; patients who are unable to walk because of paralysis, but who are up in a wheelchair will be considered ambulatory for the purpose of assessing the performance score; life expectancy must be >= 2 months for all patients
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Chemotherapy and/or biologics: Must not have received treatment within 3 weeks of entry onto this study (4 weeks if prior nitrosureas
  * Radiation: At least 4 weeks since last dose of radiation therapy to at least one lesion being used as criteria for study eligibility; only 2 weeks must elapse since the last dose of radiation (small port) to a lesion not used for study eligibility; at least 6 months must have elapsed since the last dose of prior craniospinal XRT and radiation to >= 50% of the pelvis or TBI
  * Stem Cell Transplant (SCT): >= 9 months must have elapsed since autologous hematopoietic stem cell transplant (aHSCT)
  * Prior MIBG therapy: At least 12 weeks must have elapsed since treatment with therapeutic doses of MIBG
  * Study specific limitations on prior therapy: patients who have a history of allogeneic HSCT are not eligible
* Growth factor(s): At least 7 days since the last dose of any myeloid growth factor was given
* Any patient considered for this protocol must meet the following criteria for minimum number of autologous stem cells sufficient to rescue hematopoiesis; a combination of products may be used to meet this requirement
* All stem cell products infused on this protocol must meet the following criteria for tumor analysis: No tumor cells detectable by immunocytology OR for patients who had a PBSC collection done previously and no immunocytological testing was done on the product at the time of collection: This product may be used for infusion on this study if the patient's bilateral bone marrow aspirate and biopsy specimens can be shown to be tumor free by standard histology within 4 weeks of PBSC collection
* Glomerular filtration rate (GFR) using blood draw method or 12 hour urine collection for creatinine clearance >= 100 ml/min/1.73 m^2
* Serum creatinine =< 1.5 x upper limit of normal for age
* Normal ejection fraction (>= 55%) documented by echocardiogram or radionuclide MUGA evaluation OR normal fractional shortening (>= 27%) documented by echocardiogram
* Total bilirubin < 1.5 x upper limit of normal
* AST/ALT =< 3 x upper limit of normal
* Platelets >= 75,000/uL (transfusion independent)
* Hemoglobin >= 8 g/dl (transfusion allowed)
* Because evaluation of hematopoietic toxicity is essential to this study, the same criteria will be applied to patients with tumor infiltration of the bone marrow
* Normal lung function as manifested by no dyspnea at rest and no oxygen requirement

Exclusion Criteria:

* No patients who are pregnant or lactating will be allowed to enter on study; pregnancy tests must be obtained in females who are post-menarchal; males and females of reproductive potential may not participate unless they have agreed to use an effective method of contraception while receiving therapy
* Patients with active infections requiring intravenous antivirals, antibiotics, or antifungals; patients on prolonged antifungal therapy are still eligible if they are culture negative and biopsy negative in suspected residual radiographic lesions and they meet other organ function criteria; patients who are known HIV seropositive with stable disease and lack of major health problems who are not on anti-retroviral therapy, may be eligible at the discretion of the Study Chair
* Prior treatment with Pyrazoloacridine (PZA)
* Prior history of allogeneic HSCT
* Neurologic Exclusions:

  * Acute or chronic CNS disease
  * History of seizures
  * History of cerebral bleeding or stroke
  * CNS parenchymal metastases as documented by head CT with contrast or head MRI with gadolinium performed within 30 days of study entry. Patients with epidural metastases causing mass effect on the brain are also excluded (skull metastases are allowed provided they are not associated with intracranial disease compressing or displacing the brain

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2002-12; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by dose-limiting toxicities by NCI Common Toxicity Criteria | 28 days

SECONDARY OUTCOMES:
Time to engraftment (hematopoietic recovery) | Up to 4 years
  Will be summarized with tables and with Kaplan-Meier plots.
Response by RECIST or MIBG-scans | 28 days
Survival | Up to 4 years
Time to progression | Up to 4 years
Time to failure | Time from start of treatment until death for any cause or disease progression, assessed up to 4 years
Pharmacokinetic (such as AUC, Cmax, Tmax, and clearance in the plasma) determinations | 3, 24, 72,and 192 hours after starting infusion
  Will be summarized by dose level with simple summary statistics: means (possibly after transformation) or medians, ranges, and standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Butturini, Principal Investigator — New Approaches to Neuroblastoma Treatment (NANT)
Locations (1):
- New Approaches to Neuroblastoma Treatment (NANT), Los Angeles, California, United States